CLINICAL TRIAL: NCT00713297
Title: Implementation of a Novel Computerized Physician Order Entry System to Reduce Medication Errors
Brief Title: Implementation of a Novel Computerized Physician Order Entry System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Wu, Fe-Lin, Lin/Director, Department of Pharmacy, N.T.U.H.
Other Study IDs: 200803060R
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2008-06

CONDITIONS: Computerized Physician Order Entry
Keywords: medication errors; computerized physician order entry; pharmaceutical care; chemotherapeutic agents; reengineering
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Those who will use the new CPOE system
  Interventions: Behavioral: satisfaction questionnaire

INTERVENTIONS:
Behavioral: satisfaction questionnaire — Satisfaction questionnaire
  Other Names: questionnaire

SUMMARY:
The objective of this prospective study is to build a real-time interactive platform where doctors and pharmacists may communicate and solve patients' drug-related problems (DRP) immediately and document accordingly. This study will also design a computerized physician order entry (CPOE) system utilizing default protocol for chemotherapy order entry.

DETAILED DESCRIPTION:
To err is human. Most errors are caused by problems in the system. Punishing health personnel cannot prevent the same mistakes. The only solution is a good medication system. CPOE system can prevent prescribing errors. The CPOE system is always the major step in some studies concerning reducing prescribing errors, dispensing errors or administering errors. In this user-friendly and convenient era, improvement in the CPOE system is an immediate need.

ELIGIBILITY:
Inclusion Criteria:

* NTUH pharmacists

Exclusion Criteria:

* NTUH pharmacists who have never recorded drug related problems

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NTUH pharmacists
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
the timeliness and efficiency of pharmacist's response in DRPs, the average prescription error rate and the satisfaction questionnaire before and after implementation of the new CPOE system. | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Fe-Lin L. Wu, MSCP,Ph D, Principal Investigator — Department of Pharmacy, N.T.U.H.
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan